CLINICAL TRIAL: NCT00521729
Title: Thyroid Hormones Homeostasis and Energy Metabolism Changes During Exposure to Cold Temperature in Humans
Brief Title: Metabolism and Thyroid Hormone Changes During Exposure to Cold Temperatures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Other
Other Study IDs: 070202; 07-DK-0202
Record Dates: First submitted 2007-08-25; First posted 2007-08-28 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-06-26

CONDITIONS: Obesity
Keywords: Thyroid; Thermoregulation; Catecholamines; Energy Expenditure; Obesity; Healthy Volunteer; HV
MeSH Terms: conditions — Obesity; Thyroid Diseases

INTERVENTIONS:
Procedure: Exposure to Cold Temperature

SUMMARY:
This study will examine how body metabolism adjusts to small changes in environmental temperature and how it may be related to weight loss.

Healthy, non-obese individuals between 18 and 60 years of age may be eligible for this study. The study consists of one screening visit and one 5-day admission to the NIH Clinical Center for the following procedures:

Diet: Participants follow a proscribed diet consisting of 50% carbohydrates, 20% protein and 30% fat.

DEXA scan to measure body fat. Subjects lie on a table above a source of X-rays while a very small dose of X-rays is passed through the body.

Air displacement plethysmography (Bod-Pod) to study fat composition: Subjects sit in a small booth for 10 minutes wearing a swim suit and breathing normally through a tube. This test measures the person s weight and volume precisely.

Metabolic room: Subjects stay 12 hours in a specialized room designed to measure the amount of oxygen breathed in and the amount of carbon dioxide breathed out. The room contains a private toilet and sink, treadmill, bed, desk, window, telephone and computer with television and internet access. While in this room, subjects undergo the following:

* Continuous heart rate monitor: Subjects wear an EKG monitor to analyze heart rate variability.
* Spontaneous movements: Subjects wear portable accelerometers at the hip and wrist to measure spontaneous physical movements.
* Continuous temperature monitor: Subjects swallow a small capsule that transmits internal body temperature via miniature, wireless sensors. Adhesive patches placed on the skin monitor external body temperature.
* Blood and urine collections: Subjects collect all of their urine during the 12 hours they are in the metabolic room. Blood samples are taken at specified intervals through a catheter that has been placed in a vein.
* Microdialysis: A small needle is placed into fat tissue just under the skin on the abdomen. A solution containing a minimal amount of ethanol is infused and samples of fluid are collected every 20 minutes as it leaves the fat pad. This helps determine the metabolism level. This procedure starts 30 minutes before entering the metabolic room and continues until the subject leaves the room.

Fat tissue biopsy: A small piece of fat tissue is withdrawn through a needle from under the skin on the abdomen. The sample is used to study fat tissue size and ability to store sugar.

DETAILED DESCRIPTION:
Thyroid hormones play an important role in the modulation of energy metabolism by regulating the rate of thermogenesis, i.e. the amount of heat produced to maintain the stable core temperature of the organism. Clinically, hypo- and hyperthyroidism are associated with major changes of thermoregulation and energy expenditure. While in rodents the ability of thyroid hormones in regulating the temperature and energy expenditure in response to changes of temperature is well known, its actual role in humans is poorly understood. We hypothesize that humans will respond to exposure to moderate cold by increasing the energy expenditure mediated by the thyroid hormones action and, at the same time, by decreasing the heat dispersion. This randomized, cross-over study is aimed to analyze the changes in the thyroid hormones, energy expenditure and stress hormones in response to exposure to mild changes in environmental temperature.

A total of 230 lean and overweight volunteers who are 18 years of age or older, following a two-day period of standardized diet, will be randomized to either a normal (75 (Infinite)F/24 (Infinite)C) or low-temperature (64 (Infinite)F/18 (Infinite)C) 12- or 24-hour stay in a temperature-controlled metabolic chamber. A standard meal will be provided after six hours of recording in studies performed during the daytime. After a two-day resting period the test will be then repeated at the second temperature. In order to visualize and quantify the metabolic activity of brown adipose tissue (BAT), twenty five lean study volunteers younger than 60 will be asked to undergo a 18-fluoro-deoxy-glucose PET-scan after each of the two 12-hour overnight stays in the metabolic chamber. In order to determine the impact of mitochondrial function on cold-stimulated BAT activity, a sub-group of volunteers who carry a mutation in the mitochondrial genes, succinate dehydrogenases, and age- and gender-matched control subjects, will undergo PET/CT scanning at the end of a 24-hour stay in the metabolic chamber at 18 (Infinite)C and 24 (Infinite)C.

The following parameters will be recorded and analyzed: Changes in skin and core temperature, heart rate and its variability, energy expenditure, changes in circulating thyroid hormones, ACTH, cortisol, and catecholamines. Changes in glucose uptake in relation to changes in energy expenditure will be measured by PET-scan.

The adipose tissue metabolism will be analyzed by microdialysis and study volunteers will be asked to undergo subcutaneous adipose tissue needle biopsy.

The data gathered from this study will provide a comprehensive insight into the mechanism(s) regulating the energy metabolism in response to mild cold. The results obtained from the proposed experiments might lead to the characterization of a population of subjects who are requiring excessive energy expenditure to prevent hypothermia upon cold exposure. Thus, we hypothesize that in a subset of subjects an exposure to mild cold will produce a negative energy balance ultimately facilitating weight loss.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to18
* Written informed consent
* (for SDH study only: <60 years old, documented SDH mutation without clinical evidence of pheochromocytoma or biochemical evidence of excess of catecholamines. The assessment will be performed within the context of the 00-CH-0093 protocol, P.I. Karel Pacak).

EXCLUSION CRITERIA:

* Hypo- or hyper-thyroid (history or TSH greater than 5.0 and less than 0.4 miU/L)
* Blood pressure greater than 140/90 mmHg or current antihypertensive therapy
* History of cardiovascular disease
* BMI less than or equal to 20 or greater than or equal to 35 Kg/m(2)

Diabetes mellitus (fasting serum glucose X greater than 126 mg/dL)

* Hypercholesterolemia (serum levels greater than or equal to 240 mg/dL), hypertriglyceridemia (plasma levels greater than or equal to 220 mg/dL) and/or use of antilipemic therapy
* Liver disease or ALT serum level greater than two fold the upper laboratory reference limit
* Iron deficiency (Ferritin less than 40 ng/mL males, and less than 20 ng/mL females)
* Renal insufficiency or estimated creatinine clearance less than or equal to 50 mL/min (MDRD equation)
* Claustrophobia
* History of illicit drug or alcohol abuse within the last 5 years; current use of drugs (by history) or alcohol (CAGE greater than 3)
* Psychiatric conditions or behavior that would be incompatible with safe and successful participation in this study
* Current use of medications/dietary supplements/alternative therapies known to alter thyroid function
* Current use of antiplatelet or anticoagulants
* Allergy to lidocaine
* Pregnancy/breastfeeding/hormonal contraception and childbirth within the last 24 months
* Perimenopausal (as self-described within two years from onset of amenorrhea or current complaints of hot flashes)
* Current smoker or user of tobacco products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2007-08-24; Primary Completion 2015-01-12 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in energy expenditure and in thyroid hormone levels

SECONDARY OUTCOMES:
Changes in spontaneous physical activity and in thermic effect of food

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hill JO. Understanding and addressing the epidemic of obesity: an energy balance perspective. Endocr Rev. 2006 Dec;27(7):750-61. doi: 10.1210/er.2006-0032. Epub 2006 Nov 22. PMID 17122359
- [Background] Rosen ED, Spiegelman BM. Adipocytes as regulators of energy balance and glucose homeostasis. Nature. 2006 Dec 14;444(7121):847-53. doi: 10.1038/nature05483. PMID 17167472
- [Background] Katzmarzyk PT, Leonard WR. Climatic influences on human body size and proportions: ecological adaptations and secular trends. Am J Phys Anthropol. 1998 Aug;106(4):483-503. doi: 10.1002/(SICI)1096-8644(199808)106:43.0.CO;2-K. PMID 9712477
- [Derived] Celi FS, Brychta RJ, Linderman JD, Butler PW, Alberobello AT, Smith S, Courville AB, Lai EW, Costello R, Skarulis MC, Csako G, Remaley A, Pacak K, Chen KY. Minimal changes in environmental temperature result in a significant increase in energy expenditure and changes in the hormonal homeostasis in healthy adults. Eur J Endocrinol. 2010 Dec;163(6):863-72. doi: 10.1530/EJE-10-0627. Epub 2010 Sep 8. PMID 20826525